CLINICAL TRIAL: NCT06716021
Title: Multi-Center, Placebo-Controlled, Phase 3 Study of Etripamil Nasal Spray (NS) in Patients With Atrial Fibrillation and Rapid Ventricular Rate (RVR)
Brief Title: ReVeRA-301: Etripamil in Atrial Fibrillation Phase 3
Acronym: ReVeRA-301
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Milestone Pharmaceuticals Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSP-2017-5002
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Rapid Ventricular Rate; Rapid Ventricular Response; Ventricular Rate Control
MeSH Terms: conditions — Atrial Fibrillation | interventions — etripamil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients will self-administer an initial dose of placebo for a perceived episode of AF with RVR, followed by an optional second dose 10 minutes later if symptoms persist.
  Interventions: Drug: Placebo
- Etripamil (Experimental): Patients will self-administer an initial dose of etripamil for a perceived episode of AF with RVR, followed by an optional second dose 10 minutes later if symptoms persist.
  Interventions: Drug: Etripamil

INTERVENTIONS:
Drug: Placebo — The formulation of placebo will consist of water, sodium acetate, disodium EDTA, and sulfuric acid to reproduce the same pH as the etripamil formulation.
  Arms: Placebo
Drug: Etripamil — The formulation of etripamil is for IN administration and will consist of etripamil, water, acetic acid, disodium ethylene-diamine-tetra-acetic acid (EDTA), and sulfuric acid. The dose of etripamil to be evaluated in this study is 70 mg with an optional second dose of 70 mg 10 minutes after the first dose if symptoms persist.
  Other Names: MSP-2017
  Arms: Etripamil

SUMMARY:
This is a multi-national, multi-center, randomized, double-blind, placebo-controlled study to evaluate the effects of etripamil NS in patients with atrial fibrillation (AF). This study includes Screening Visit, Randomization Visit, a Treatment Period with scheduled Follow-up Visits (Monthly Follow-up and Post-treatment Follow-up Visits), a Final Study Visit, and an End of Study Telephone Follow up Visit.

Each patient will be randomized 1:1 to receive placebo or 70 mg Etripamil NS regimens. Patients will self-administer study drug for a perceived episode of AF with RVR with an initial dose of placebo or 70 mg etripamil NS, followed by an optional second dose of the same study drug 10 minutes after the first dose if the patient continues to experience symptoms. Patients may treat up to a maximum of 4 episodes in the study.

Informed consent will be obtained prior to any study procedures.

DETAILED DESCRIPTION:
This is a multi-national, multi-center, randomized, double-blind, placebo-controlled study to evaluate the effects of etripamil NS in patients with AF. This study includes a Screening Visit, Randomization Visit, Treatment Period with Follow-up Visits (Monthly Follow-up Visits, and Post-treatment Follow-up Visits), a Final Study Visit, and an End of Study Telephone Follow-up Visit.

Each patient will be randomized in a 1:1 ratio to receive Placebo or 70 mg Etripamil NS regimens. Patients will self-administer study drug for a perceived episode of AF with RVR as follows: an initial dose of placebo or 70 mg etripamil NS, followed by an optional second dose 10 minutes after the first dose if the patient continues to experience symptoms.

Patients may treat up to a maximum of 4 episodes in the study. Informed consent must be obtained prior to any study procedures.

Screening Visit:

Patients with a history of symptomatic AF with RVR will be selected by the Investigator. The screening procedures will include obtaining informed consent, a review of inclusion/exclusion criteria, vital signs, a physical examination, measuring height and weight, screening lab tests, 12-lead electrocardiogram (ECG), recording demographics and medical history and recording of any concomitant medications.

Documentation of AF with RVR, and other data if relevant or requested (e.g. concomitant medications, medical history) will be submitted for Sponsor medical review to confirm and approve patient eligibility for randomization.

Randomization Visit:

Patients eligible for randomization will return to the site to confirm eligibility, record any changes in concomitant medications and adverse events (AEs), and receive training in study procedures including recognizing the presence of customary symptoms of AF, use of the ECG cardiac monitoring system (CMS) device, and electronic patient reported outcome (ePRO) device. Patients will then be randomized 1:1 to placebo or etripamil NS and dispensed study drug kits.

Treatment Period:

When randomized patients identify symptoms of an episode of AF with RVR, they will perform a sequence of steps, including affixing an ECG CMS device, confirming they have an elevated ventricular rate (≥110 bpm), self-administering study drug, and completing an ePRO at specified times post-study drug. A caregiver may help the patient with these procedures. Administration of the study drug regimen during an AF episode is as follows: an initial dose of study drug followed by an optional second dose 10 minutes after the first dose if symptoms persist.

Patients should refrain from additional treatment for their AF with RVR until 45 minutes after their first dose of study drug, after which they should treat their episode as needed per physician-recommended standards of care.

A patient may treat up to 4 episodes during the study.

Follow-up Visits:

Monthly Follow-up Visits Follow-up Visits will occur approximately monthly from the time of randomization until the patient completes the study. These visits will be conducted via site visit or telephone. AEs and concomitant medications therapies will be collected and recorded, continued patient eligibility will be assessed based on information collected, and any re-training on study procedures will be conducted.

Post-treatment Follow-up Visit(s) A Post-treatment Follow-up Visit will occur at the study site within 14 days after a patient administers study drug during the Treatment Period. Up to 4 treated episodes of perceived AF are allowed per patient. AEs and concomitant medications will be collected and recorded, weight and vital signs will be measured, the CMS report from the treated episode will be reviewed, patient eligibility confirmed, study drug kits will be collected for drug accountability, and if applicable the patient will be re-randomized and additional study drug kits dispensed. A focused physical examination will also be performed if needed to assist in the evaluation of any reported AEs.

Details on any medical interventions (e.g. oral medication, intravenous [IV] medication, visits to the emergency department or health-care facility, and/or arrhythmia-related procedure [such as cardioversion]) associated with the treated episode will be collected.

If a patient has completed or will not be continuing in the study, Final Study Visit procedures will be performed.

Final Study Visit:

A Final Study Visit will occur at the study site after a patient administers study drug for the final time during the Treatment Period, or if the patient has completed participation in the study for any other reason. This Visit may be conducted at the same time as a Post-treatment Follow-up Visit.

AEs and concomitant medications will be collected and recorded, weight and vital signs will be measured, the CMS report from the treated episode will be reviewed. A focused physical examination will also be performed if needed to assist in the evaluation of any reported AEs. Reasons for study completion or withdrawal will be collected, and the patient will return the ECG monitoring device and ePRO device at this visit. Study drug kits, ECG CMS devices, and ePRO will be collected.

End of Study Telephone Follow-Up Visit:

An End of Study Telephone Follow-Up Visit will be completed approximately 30 days after the Final Study Visit to follow-up on any ongoing AEs. This visit is not required for patients who did not use the study drug within 30 days before their Final Study Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and over.
2. Provision of written informed consent.
3. Documented history of symptomatic AF (paroxysmal, persistent, or permanent) with a ventricular rate of ≥110 bpm.

   * Documentation: electrocardiogram (ECG) tracing (including 12-lead ECG or ECG strip) showing AF with ventricular rate ≥110 beats per minute (bpm). This ECG documentation (anonymized with study Patient ID only) will be submitted to the Sponsor after screening and prior to randomization to confirm diagnosis of AF with RVR and eligibility to be randomized in the study. Patients who have undergone a prior ablation procedure for AF or for an AF-trigger must have documented AF with RVR post-ablation for study eligibility.
4. Documented history of repeated (at least 2 within the prior 12 months) and prolonged (at least 20 minutes) symptomatic episodes of AF with elevated (perceived or measured) heart rate (HR).

   * Documentation: Patient description, other history, or medical records. Patients who have undergone a prior ablation procedure for AF or for an AF-trigger must fulfill this criterion post-ablation for study eligibility.
5. Receiving appropriate antithrombotic/anticoagulation therapy as per applicable national and/or local guidelines for AF management.
6. Women of childbearing potential must have a negative pregnancy test at Screening and agree to use at least 1 highly effective form of contraception from time of randomization until 7 days after the last administration of study drug and must be willing to discontinue from the study should they become or plan to become pregnant.

Exclusion Criteria:

1. Patients with a primary diagnosis of atrial flutter (typical or atypical) or atrial tachycardia. Patients with AF who have been observed to also experience atrial flutter within the same episode (i.e., "AFib/Flutter" or an admixture of AF and flutter within the same episode) are eligible.
2. History of any of the following within the last 6 months: Class 3 or 4 angina per Canadian Cardiovascular Society (CCS) criteria; ischemic chest pain during AF episodes; acute coronary syndrome, unless the patient has been successfully revascularized; coronary artery bypass grafting or open-chest valve surgery.
3. History of heart failure (HF) New York Heart Association (NYHA) classification ≥Class III within the last 3 months.

   * The etiology of any HF should have been previously evaluated and addressed.
   * HF with a reduced ejection fraction and/or HF with a preserved ejection fraction are acceptable.
4. History of hemodynamic instability during AF, i.e., symptoms or signs of severe hypotension, or syncope due to a pause upon conversion from AF to sinus rhythm (SR).
5. History of unexplained syncope.
6. History of, or ECG evidence at the screening visit, of: sick sinus syndrome, Mobitz II second- or third-degree atrioventricular (AV) block bradycardia (<40 bpm) or pauses >3 seconds during waking hours, without a pacemaker.
7. History of, or ECG evidence at the Screening visit, of: torsades de pointes, ventricular fibrillation, or ventricular tachycardia, Brugada syndrome, an antegrade conducting accessory bypass tract (e.g., Wolff-Parkinson-White or Lown-Ganong-Levine syndromes), or long QT syndrome.
8. History of stroke, transient ischemic attack or peripheral embolism within the last 3 months.
9. CHA2DS2-VASc score of >5.
10. Planned AF or AV node ablation within the next 3 months.
11. Uncorrected, severe aortic or mitral stenosis.
12. Hypertrophic cardiomyopathy with outflow tract obstruction.
13. History of sensitivity to verapamil or to any components of the investigational product.
14. History of recent or current chronic alcohol or drug abuse that, in the opinion of the Investigator, could impact the validity of the study results.
15. Currently participating in another drug or device study, or has received an investigational drug or device within 30 days prior to Screening.
16. Any other significant co-morbid condition that may negatively impact the patient's participation in the study or likely result in non-compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the efficacy of etripamil NS over placebo in patients with AF. | 30 minutes from first drug administration
  The maximum reduction in ventricular rate, measured from ECG CMS recordings, within 30 minutes from first drug administration

CONTACTS AND LOCATIONS:
Overall Officials: James E. Ip, MD, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: No